CLINICAL TRIAL: NCT05850208
Title: A Randomized, Open and Routine Parallel Controlled Clinical Study on the Safety and Efficacy of Autologous Bone Marrow Mesenchymal Stem Cells (BMSCs) Transplantation in the Treatment of Ischemic Stroke
Brief Title: Autologous Bone Marrow Mesenchymal Stem Cells (BMSCs) Transplantation in the Treatment of Ischemic Stroke
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJYY.ZTGSJCZGXB-HBT-V2.3-CTP
Record Dates: First submitted 2022-08-24; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine treatment group (No Intervention): No special measures were taken and routine treatment was adopted
- BMSCs group (Experimental): BMSCs were transplanted on the basis of routine treatment: the transplanted cells were injected intravenously and transplanted in two times at a dose of 1 × 106/kg body weight, each volume was 80ml ± 5ml, and the time interval between two transplants was 1 week
  Interventions: Biological: Transplantation of self BMSCs

INTERVENTIONS:
Biological: Transplantation of self BMSCs — Bone marrow was collected, cultured in vitro and injected back into the body
  Arms: BMSCs group

SUMMARY:
This study is to evaluated the safety and efficacy of BMSCs transplantation in the treatment of ischemic stroke, so as to provide a basis for future clinical application of BMSCs transplantation in the treatment of ischemic stroke.

DETAILED DESCRIPTION:
1. Routine treatment:

   1.1. If arterial plaque is found, use lipid-lowering therapy (routine dose of atorvastatin or rosuvastatin). If no plaque is found, use atorvastatin or rosuvastatin based on the maintenance of normal blood lipid;

   1.2. If venous thrombosis or arterial plaques are found in the lower limbs, use dabigatran to prevent platelet aggregation; if no vascular problems are found in the lower limbs, use aspirin or clopidogrel to prevent platelet aggregation;

   1.3. During the treatment, cerebrovascular stenosis (non responsible vessels) can be treated intravascularly;

   1.4. The use of neurotrophic drugs is prohibited during the study;

   1.5. Elevated homocysteine was treated with mecobalamin and folic acid;

   1.6. Hypertension, diabetes and other basic diseases receive routine treatment, and the combined medication is recorded in the case report form.
2. Grouping:

2.1. BMSCs group: BMSCs were transplanted on the basis of routine treatment: the transplanted cells were injected intravenously and transplanted in two times, with a dose of 1 × 106 / kg body weight, each volume of 80ml ± 5ml, and the time interval between two transplants was 1 week;

2.2. Routine treatment group: only receiving routine treatment;

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-65 years old in the rehabilitation period of cerebral infarction (including subacute stage, chronic stage and sequelae stage, with onset time ≤ 3 years), regardless of gender;
2. Definite cerebral infarction in the blood supply area of middle cerebral artery confirmed by imaging;
3. There are clear neurological deficits, such as motor and cognitive dysfunction (National Institutes of Health Stroke Scale 7 < NIHSS < 21 points);
4. Those who agree to take effective contraceptive measures during the study period, and women of childbearing age have negative pregnancy test;
5. Sign the informed consent of the patient and agree to participate in all visits, examinations and treatments as required by the study protocol.

Exclusion Criteria:

1. Lacunar cerebral infarction;
2. Acute cerebral infarction, onset time < 2 weeks;
3. Mild ischemic stroke or mild neurological impairment or severe ischemic stroke, with coma;
4. Patients with moyamoya disease, vascular malformation, hemangioma and carotid stenosis exceeding 70%;
5. Patients with severe heart valve disease or confirmed intractable atrial fibrillation;
6. Complicated with intracranial hemorrhage or tumor;
7. Patients with cerebral infarction caused by blood system diseases, or those with previous blood history or family history of blood diseases;
8. Any one of 5 items of hepatitis B virus (HBsAg, HBsAb, HBeAg, HBeAb, HBcAb), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody and syphilis spiral physical examination;
9. Those with severe respiratory or circulatory system or liver and kidney dysfunction who cannot tolerate treatment and examination;
10. Severe febrile disease or viral disease in the past 12 weeks;
11. Malignant tumor;
12. Those who have a previous history of autoimmune diseases or a family history of autoimmune diseases;
13. Previous history of drug allergy;
14. Pregnant or lactating women;
15. Those who are participating or have participated in this study or participated in other clinical trials within 12 weeks before enrollment;
16. Other circumstances that the investigator considers inappropriate for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference in National Institutes of Health Stroke Scale (NIHSS) score from baseline after the first transplant. | 96 weeks ±30 days after the first transplantation
  The difference in National Institutes of Health Stroke Scale (NIHSS) score from baseline at week 96 ±30 days after the first transplant.

SECONDARY OUTCOMES:
The difference from baseline in National Institutes of Health Stroke Scale (NIHSS) score after the first transplantation | 48 weeks ±15 days after the first transplantation
  The difference from baseline in National Institutes of Health Stroke Scale (NIHSS) score at 48 weeks ±15 days after the first transplantation
Improvement rate of the modified Barthel Index Rating Scale score from baseline after the first transplant | 48 weeks ±15 days after the first transplantation
  Improvement rate of the modified Barthel Index Rating Scale score from baseline at 48 weeks ±15 days after the first transplantation
Improvement rate of the modified Barthel Index Rating Scale score from baseline | 96 weeks ±30 days after the first transplantation
  Improvement rate of the modified Barthel Index Rating Scale score from baseline at 96 weeks ±30 days after the first transplant
Improvement rate of Fugl-Meyer scale score from baseline after the first transplantation | 48 weeks ±15 days after the first transplantation
  Improvement rate of Fugl-Meyer scale score from baseline at 48 weeks ±15 days after the first transplantation
Improvement rate of Fugl-Meyer scale score from baseline after the first transplantation | 96 weeks ±30 days after the first transplantation
  Improvement rate of Fugl-Meyer scale score from baseline at 96 weeks ±30 days after the first transplantation
Improvement rate of Simple Mental State Examination Scale (MMSE) score | 48 weeks ±15 days after the first transplantation
  Improvement rate of Simple Mental State Examination Scale (MMSE) score from baseline at 48 weeks ±15 days after the first transplantation
Improvement rate of Simple Mental State Examination Scale (MMSE) score | 96 weeks ±30 days after the first transplantation
  Improvement rate of Simple Mental State Examination Scale (MMSE) score from baseline at 96 weeks ±30 days after the first transplantation
The time course of the left abductor pollicis brevis and right abductor pollicis brevis of the motor evoked potential decreased from baseline after the first transplantation | 48 weeks ±15 days after the first transplantation
  The time course of the left abductor pollicis brevis and right abductor pollicis brevis of the motor evoked potential decreased from baseline at 48 weeks ±15 days after the first transplantation
The time course of the left abductor pollicis brevis and right abductor pollicis brevis of the motor evoked potential decreased from baseline after the first transplantation | 96 weeks ±30 days after the first transplantation
  The time course of the left abductor pollicis brevis and right abductor pollicis brevis of the motor evoked potential decreased from baseline at 96 weeks ±30 days after the first transplantation
MT increase rate from baseline in the left abductor Pollicis brevis and right abductor pollicis brevis of the motor evoked potential after the first transplantation | 48 weeks ±15 days after the first transplantation
  MT increase rate from baseline in the left abductor Pollicis brevis and right abductor pollicis brevis of the motor evoked potential at 48 weeks ±15 days after the first transplantation
MT increase rate from baseline in the left abductor Pollicis brevis and right abductor pollicis brevis of the motor evoked potential after the first transplantation | 96 weeks ±30 days after the first transplantation
  MT increase rate from baseline in the left abductor Pollicis brevis and right abductor pollicis brevis of the motor evoked potential at 96 weeks ±30 days after the first transplantation
The time course of the upper limb sensory evoked potential N9(left), N11(left), N20(left), N9(right), N11(right), N20(right) decreased from baseline after the first transplantation | 48 weeks ±15 days after the first transplantation
  The time course of the upper limb sensory evoked potential N9(left), N11(left), N20(left), N9(right), N11(right), N20(right) decreased from baseline at 48 weeks ±15 days after the first transplantation
The time course of the upper limb sensory evoked potential N9(left), N11(left), N20(left), N9(right), N11(right), N20(right) decreased from baseline after the first transplantation | 96 weeks ±30 days after the first transplantation
  The time course of the upper limb sensory evoked potential N9(left), N11(left), N20(left), N9(right), N11(right), N20(right) decreased from baseline at 96 weeks ±30 days after the first transplantation
Rate of increase from baseline amplitude of the upper limb sensory evoked potential N9(left), N11(left), N20(left), N9(right), N11(right), N20(right) after the first transplantation | 48 weeks ±15 days after the first transplantation
  Rate of increase from baseline amplitude of the upper limb sensory evoked potential N9(left), N11(left), N20(left), N9(right), N11(right), N20(right) at 48 weeks ±15 days after the first transplantation
Rate of increase from baseline amplitude of the upper limb sensory evoked potential N9(left), N11(left), N20(left), N9(right), N11(right), N20(right) after the first transplantation | 96 weeks ±30 days after the first transplantation
  Rate of increase from baseline amplitude of the upper limb sensory evoked potential N9(left), N11(left), N20(left), N9(right), N11(right), N20(right) at 96 weeks ±30 days after the first transplantation
Changes in CTA from baseline after the first transplantation | 48 weeks ±15 days after the first transplantation
  Changes in CTA from baseline at 48 weeks ±15 days after the first transplantation
Changes in CTA from baseline after the first transplantation | 96 weeks ±30 days after the first transplantation
  Changes in CTA from baseline at 96 weeks ±30 days after the first transplantation
Changes in CTP from baseline after the first transplantation | 96 weeks ±30 days after the first transplantation
  Changes in CTP from baseline at 96 weeks ±30 days after the first transplantation
Changes in CTP from baseline after the first transplantation | 48 weeks ±15 days after the first transplantation
  Changes in CTP from baseline at 48 weeks ±15 days after the first transplantation
Changes in mRS Scores from baseline after the first transplantation | 48 weeks ±15 days after the first transplantation
  Changes in mRS Scores from baseline at 48 weeks ±15 days after the first transplantation
Changes in mRS Scores from baseline after the first transplantation | 96 weeks ±30 days after the first transplantation
  Changes in mRS Scores from baseline at 96 weeks ±30 days after the first transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Not yet determined